CLINICAL TRIAL: NCT03024892
Title: Intra-gallbladder or Systemic Indocyanide Green Injection Facilitate Cholecystectomy in Acute Cholecystitis , Gallstone and Gallbladder Polyp Patients.
Brief Title: Intra-gallbladder or Systemic Indocyanide Green Injection Facilitate Cholecystectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGMH-IRB-104-5333A3
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Fluorenscent Image Guided Surgery; Indocyanide Green
Keywords: Fluorenscent image guided surgery; indocyanide green; laparoscopic cholecystectomy; common bile duct injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ICG gallbladder (Experimental): patients who received ICG injection via gallbladder and received fluroscence image guided surgery
  Interventions: Procedure: ICG GB
- ICG IV (Experimental): patients who received ICG injection via peripheral vein and received fluroscence image guided surgery
  Interventions: Procedure: ICG IV
- LC conventional (Sham Comparator): Patients received conventional laparoscopic cholecystectomy
  Interventions: Procedure: LC conventional
- LC conventional and IOC (Sham Comparator): Patients received conventional laparoscopic cholecystectomy + intraoperative cholangiography
  Interventions: Procedure: LC conventional and IOC

INTERVENTIONS:
Procedure: ICG GB — ICG was given by intra-gallbladder injection, then the near-infrared image guide laparoscopic cholecystectomy were performed.
  Arms: ICG gallbladder
Procedure: ICG IV — ICG was given by systemic injection, then the near-infrared image guide laparoscopic cholecystectomy were performed.
  Arms: ICG IV
Procedure: LC conventional — simple laparoscopic cholecystectomy was performed under white light image.
  Arms: LC conventional
Procedure: LC conventional and IOC — simple laparoscopic cholecystectomy was performed under white light image and intraoperaitve cholangiography guidance.
  Arms: LC conventional and IOC

SUMMARY:
The investigators will collect the pre-operative medical history and arrange physical examination, life quality evaluation, blood and biochemical test. The Patients with acute cholecytitis, gallstone or gallbladder polyp without interventional treatment or cholecystitis after percurtaneus gallbladder drainage(PTGBD) were involved in this study. Four laparoscopic ports were introduced and the pneumoperitoneum (12mmHg) was established. In study group , ICG was give by intra-gallbladder injection or systemic injection, the cholecystectomy were performed . In control group, no ICG was given and traditional cholecystectomy were performed. A near-infrared optimized laparoscope was used to detect the ICG fluorescence signal arising from gallbladder , cystic duct and common bile duct before cholecystectomy in study group. According to the enhancement of ICG, the cholecystectomy was started from cystic duct in Calot's triangle.Time to gallbladder removed was recorded. Conversion rate, post-operative morbidity and mortality will be recorded as well .

DETAILED DESCRIPTION:
Back Ground:

Laparoscopic cholecystectomy(LC) is the one of most common procedure done by minimal invasive surgery worldwide but the common bile duct(CBD) injury still happened even the existence of standard technique with growing experience and new technology, especial in cholecystitis. Image guided surgery created new concept for fluorescent cholangiography to demonstrate the anatomy of CBD by using indocyanine green (ICG) intravenous injection before operation to decreased complication. The result is positive but the border of gallbladder can't be seen very well in systemic injection . In cholecystitis, the border between gallbladder and common bile duct is important as well as CBD and cystic duct.

Purpose:

The investigators hypothesized injection of ICG into gallbladder directly will be helpful to identify cystic duct, CBD and the border of gallbladder as well as systemic injection . The purpose of this study was to evaluate feasibility of this image guide surgery

Study Design:

The investigators will collect the pre-operative medical history and arrange physical examination, life quality evaluation, blood and biochemical test. The Patients with acute cholecytitis, gallstone or gallbladder polyp without interventional treatment or cholecystitis after percurtaneus gallbladder drainage(PTGBD) were involved in this study. Four laparoscopic ports were introduced and the pneumoperitoneum (12mmHg) was established. In study group , ICG was give by intra-gallbladder injection or systemic injection, the cholecystectomy were performed . In control group, no ICG was given and traditional cholecystectomy were performed. A near-infrared optimized laparoscope was used to detect the ICG fluorescence signal arising from gallbladder , cystic duct and common bile duct before cholecystectomy in study group. According to the enhancement of ICG, the cholecystectomy was started from cystic duct in Calot's triangle. Time to gallbladder removed was recorded. Conversion rate, post-operative morbidity and mortality will be recorded as well . The investigators intend to collect 600 patients. 150 patients will receive ICG injection via gallbladder as image guided surgery, 150 patients will receive ICG injection via systemic injection as image guided surgery , the other 300 patients who refuse will be the control group(150 patients for LC and 150 patients for LC + intra-operative cholangiography).

Expected results A. Publish Intra-gallbladder indocyanide green injection via drainage route facilitate cholecystectomy in acute cholecystitis。 B. Publish Comparison of systemic and intra-gallbladder injection of indocyanide green in benefit for cholecystectomy C. Extend to publish Near-infrared cholangiography decreased learning curve of laparoscopic cholecystectomy for medical student D. Near- infrared laparoscope education textbook and clinical case analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute cholecytitis, gallstone or gallbladder polyp without interventional treatment or cholecystitis after percurtaneus gallbladder drainage(PTGBD) were involved in this study.

Exclusion Criteria:

* a.Pregnancy and Breast feeding female.
* b.Patients have another severe medical diseases.(ex: heart failure, respiratory failure and stroke etc.)
* c.Not suitable for patients receiving anesthesia.
* d.Alcoholism, drug abuse and psychopaths.
* e.Iodine allergies and renal failure patients.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Hartmann's pouch identification ( white light and infrared fluroscence image) | intra-operative period
  evaluation rate the visualization of Hartmann's pouch between two method
Cystic duct identification ( white light and infrared fluroscence image) | intra-operative period
  evaluation rate the visualization of Hartmann's pouch between two method
CBD identification ( white light and infrared fluroscence image) | intra-operative period
  evaluation rate the visualization of Hartmann's pouch between two method
CHD identification ( white light and infrared fluroscence image) | intra-operative period
  evaluation rate the visualization of Hartmann's pouch between two method
conversion rate | intra-operative period
  the rate for calculate the conversion from laparoscopic cholecystectomy to open cholecystectomy

SECONDARY OUTCOMES:
CBD injury | post op day 3
  evaluation of clinical S/S for jaundice , if suspect CBD injury then arrange examination
Post op morbidity | Post op day 7
  any complication related to surgery
Post op mortality | Post op day 30
  any mortality related to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Liao, MD, Principal Investigator — Chang Gung Memorial Hospital; Shang-Yu Wang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Niaosong, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Avgerinos C, Kelgiorgi D, Touloumis Z, Baltatzi L, Dervenis C. One thousand laparoscopic cholecystectomies in a single surgical unit using the "critical view of safety" technique. J Gastrointest Surg. 2009 Mar;13(3):498-503. doi: 10.1007/s11605-008-0748-8. Epub 2008 Nov 14. PMID 19009323
- [Background] Paczynski A, Koziarski T, Stanowski E, Krupa J. Extrahepatic bile duct injury during laparoscopic cholecystectomy -- own material. Med Sci Monit. 2002 Jun;8(6):CR438-40. PMID 12070436
- [Background] Shea JA, Healey MJ, Berlin JA, Clarke JR, Malet PF, Staroscik RN, Schwartz JS, Williams SV. Mortality and complications associated with laparoscopic cholecystectomy. A meta-analysis. Ann Surg. 1996 Nov;224(5):609-20. doi: 10.1097/00000658-199611000-00005. PMID 8916876
- [Background] Gutt CN, Encke J, Koninger J, Harnoss JC, Weigand K, Kipfmuller K, Schunter O, Gotze T, Golling MT, Menges M, Klar E, Feilhauer K, Zoller WG, Ridwelski K, Ackmann S, Baron A, Schon MR, Seitz HK, Daniel D, Stremmel W, Buchler MW. Acute cholecystitis: early versus delayed cholecystectomy, a multicenter randomized trial (ACDC study, NCT00447304). Ann Surg. 2013 Sep;258(3):385-93. doi: 10.1097/SLA.0b013e3182a1599b. PMID 24022431
- [Background] Zafar SN, Obirieze A, Adesibikan B, Cornwell EE 3rd, Fullum TM, Tran DD. Optimal time for early laparoscopic cholecystectomy for acute cholecystitis. JAMA Surg. 2015 Feb;150(2):129-36. doi: 10.1001/jamasurg.2014.2339. PMID 25517723
- [Background] Viste A, Jensen D, Angelsen JH, Hoem D. Percutaneous cholecystostomy in acute cholecystitis; a retrospective analysis of a large series of 104 patients. BMC Surg. 2015 Mar 8;15:17. doi: 10.1186/s12893-015-0002-8. PMID 25872885
- [Background] Suzuki K, Bower M, Cassaro S, Patel RI, Karpeh MS, Leitman IM. Tube cholecystostomy before cholecystectomy for the treatment of acute cholecystitis. JSLS. 2015 Jan-Mar;19(1):e2014.00200. doi: 10.4293/JSLS.2014.00200. PMID 25848180
- [Background] Mir IS, Mohsin M, Kirmani O, Majid T, Wani K, Hassan MU, Naqshbandi J, Maqbool M. Is intra-operative cholangiography necessary during laparoscopic cholecystectomy? A multicentre rural experience from a developing world country. World J Gastroenterol. 2007 Sep 7;13(33):4493-7. doi: 10.3748/wjg.v13.i33.4493. PMID 17724807
- [Background] Kaczynski J, Hilton J. A gallbladder with the "hidden cystic duct": A brief overview of various surgical techniques of the Calot's triangle dissection. Interv Med Appl Sci. 2015 Mar;7(1):42-5. doi: 10.1556/IMAS.7.2015.1.4. Epub 2015 Mar 20. PMID 25838927
- [Background] Sanjay P, Fulke JL, Exon DJ. 'Critical view of safety' as an alternative to routine intraoperative cholangiography during laparoscopic cholecystectomy for acute biliary pathology. J Gastrointest Surg. 2010 Aug;14(8):1280-4. doi: 10.1007/s11605-010-1251-6. Epub 2010 Jun 10. PMID 20535578
- [Background] Sanjay P, Kulli C, Polignano FM, Tait IS. Optimal surgical technique, use of intra-operative cholangiography (IOC), and management of acute gallbladder disease: the results of a nation-wide survey in the UK and Ireland. Ann R Coll Surg Engl. 2010 May;92(4):302-6. doi: 10.1308/003588410X12628812458617. PMID 20501016
- [Background] Diana M, Noll E, Diemunsch P, Dallemagne B, Benahmed MA, Agnus V, Soler L, Barry B, Namer IJ, Demartines N, Charles AL, Geny B, Marescaux J. Enhanced-reality video fluorescence: a real-time assessment of intestinal viability. Ann Surg. 2014 Apr;259(4):700-7. doi: 10.1097/SLA.0b013e31828d4ab3. PMID 23532109
- [Background] Kong SH, Noh YW, Suh YS, Park HS, Lee HJ, Kang KW, Kim HC, Lim YT, Yang HK. Evaluation of the novel near-infrared fluorescence tracers pullulan polymer nanogel and indocyanine green/gamma-glutamic acid complex for sentinel lymph node navigation surgery in large animal models. Gastric Cancer. 2015 Jan;18(1):55-64. doi: 10.1007/s10120-014-0345-3. Epub 2014 Jan 31. PMID 24481855
- [Background] Boni L, David G, Mangano A, Dionigi G, Rausei S, Spampatti S, Cassinotti E, Fingerhut A. Clinical applications of indocyanine green (ICG) enhanced fluorescence in laparoscopic surgery. Surg Endosc. 2015 Jul;29(7):2046-55. doi: 10.1007/s00464-014-3895-x. Epub 2014 Oct 11. PMID 25303914
- [Background] Ishizawa T, Bandai Y, Ijichi M, Kaneko J, Hasegawa K, Kokudo N. Fluorescent cholangiography illuminating the biliary tree during laparoscopic cholecystectomy. Br J Surg. 2010 Sep;97(9):1369-77. doi: 10.1002/bjs.7125. PMID 20623766
- [Background] Schols RM, Bouvy ND, van Dam RM, Masclee AA, Dejong CH, Stassen LP. Combined vascular and biliary fluorescence imaging in laparoscopic cholecystectomy. Surg Endosc. 2013 Dec;27(12):4511-7. doi: 10.1007/s00464-013-3100-7. Epub 2013 Jul 23. PMID 23877766
- [Background] Kilkenny C, Browne WJ, Cuthill IC, Emerson M, Altman DG. Improving bioscience research reporting: the ARRIVE guidelines for reporting animal research. PLoS Biol. 2010 Jun 29;8(6):e1000412. doi: 10.1371/journal.pbio.1000412. No abstract available. PMID 20613859
- [Background] Liu YY, Pop R, Diana M, Kong SH, Legner A, Beaujeux R, Marescaux J. Real-time fluorescence angiography by intra-arterial indocyanine green injection to identify obscure gastrointestinal bleeding territory: proof of concept in the porcine model. Surg Endosc. 2016 May;30(5):2143-50. doi: 10.1007/s00464-015-4460-y. Epub 2015 Aug 15. PMID 26275550
- [Background] Liu YY, Kong SH, Diana M, Legner A, Wu CC, Kameyama N, Dallemagne B, Marescaux J. Near-infrared cholecysto-cholangiography with indocyanine green may secure cholecystectomy in difficult clinical situations: proof of the concept in a porcine model. Surg Endosc. 2016 Sep;30(9):4115-23. doi: 10.1007/s00464-015-4608-9. Epub 2015 Oct 28. PMID 26511116